CLINICAL TRIAL: NCT06400849
Title: Comparison of the Efficacy of Cryotherapy Combined With Compression in Preventing the Development of Paclitaxel-induced Peripheral Neuropathy in Non-metastatic Breast Cancer: A Prospective, Single-centre, Self-controlled Trial
Brief Title: Comparison of the Efficacy of Cryotherapy Combined With Compression in Preventing Neuropathy
Acronym: ARIANE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/73
Record Dates: First submitted 2024-04-09; First posted 2024-05-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Non-metastatic Breast Cancer
Keywords: Non-metastatic breast cancer; Peripheral neuropathy; paclitaxel; cryotherapy; compression therapy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Open-label, single-centre, randomised (1:1), stratified, self-controlled cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy only (Active Comparator): Single group, same patient, Homolateral wearing of cryotherapy devices only on hands and feet
  Interventions: Device: cryotherapy alone of the upper or lower limbs
- Cryptherapy and compression (Experimental): Single group, same patient, Homolateral wearing of cryotherapy and compression devices on hands and feet
  Interventions: Device: cryotherapy and crompression of the upper or lower limbs

INTERVENTIONS:
Device: cryotherapy alone of the upper or lower limbs — Self-controlled trial with only standard cryotherapy. Compression glove and foot sock will only be worn on one hand and one leg on the same side allocated by randomisation
  Arms: Cryotherapy only
Device: cryotherapy and crompression of the upper or lower limbs — Self-controlled trial adding compression to standard cryotherapy. Compression glove and foot sock will only be worn on one hand and one leg on the same side allocated by randomisation
  Arms: Cryptherapy and compression

SUMMARY:
Breast cancer is the most frequently diagnosed cancer in the world. In France, 58,000 new cases were detected in 2018. Breast cancer is therefore the most common cancer in women. The 5-year survival rate for all stages combined is 88%. These excellent survival figures have been achieved thanks to improvements in treatment, including the advent of chemotherapy. The majority of patients will be cured of their cancer, so post-cancer quality of life is a major issue, hence the importance of trying to reduce long-term sequelae.

Taxanes are one of the main cytotoxic anticancer agents used in the treatment of breast cancer. However, taxanes have a direct effect on the central and peripheral nervous systems and can induce chemotherapy-induced peripheral neuropathy (CIPN). The mechanisms of NPIC by taxanes are not fully understood. CINP is manifested by symptoms of paresthesia, numbness, burning, pain, altered temperature perception, myalgia, myopathy, fine motor difficulties, gait and balance disturbances, muscle weakness in the lower limbs and/or functional decline.

NPIC occurs in 80 to 97% of patients treated with taxanes and is the main limiting toxicity during paclitaxel administration. NPIC often leads to postponement or reduction of dose, or even discontinuation of treatment. In addition, NPIC may last for several months or even years after the end of anti-cancer chemotherapy and represents the main long-term sequelae. This can promote and/or exacerbate symptoms of psychological distress (depressive symptoms and symptoms of anxiety) and lead to a reduction in quality of life (QoL). Prevention of NIPC is therefore a major issue in breast cancer treatment. According to the 2014 guidelines from the American Society of Clinical Oncology, prevention and treatment of IPN are inadequate with current weapons, and there is an urgent need to evaluate and find new methods of prevention. One of the challenges in the management of NIPC will be to reduce the pain induced without diminishing the anti-tumour effect of anti-cancer agents.

In recent years, the effectiveness of cryotherapy using a frozen glove and compression therapy using surgical gloves (SG) in preventing taxane-induced PINC has been reported. During chemotherapy, patients wore a frozen glove on one hand and two surgical gloves of the same size on the other hand continuously. Recent study explained how compression therapy and cryotherapy shared a similar mechanism of reducing drug exposure due to vasoconstriction during paclitaxel infusion. The low temperature associated with cryotherapy would reduce paclitaxel uptake and peripheral nerve damage, or mechanotransduction, and allow a reduction in NIPC.

To date, no study has investigated the efficacy of combining the two means of prevention. The current standard at the Centre Antoine Lacassagne is cryotherapy. The aim of this prospective, self-controlled trial is therefore to compare the efficacy of cryotherapy combined with compression prevention versus cryotherapy alone in preventing paclitaxel-induced peripheral neuropathy in patients undergoing adjuvant treatment for localised breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years ;
* Performance Status (PS): 0 to 2
* Women with localised or locally advanced breast cancer of any histology
* Indication for treatment with 3 to 4 cycles of paclitaxel (+/- trastuzumab, pertuzumab, carboplatin or endoxan) as adjuvant or neoadjuvant therapy. The choice of the number of cycles will be at the investigator's discretion.
* Symmetry of upper limb peripheral neuropathy grade ≤ 1 according to CTCAE version 5.0 at inclusion.
* Presence of radial pulses in the upper limbs.
* Presence of tibio-posterior and tibio-anterior ankle pulses or ankle systolic pressure index > 0.9.
* Patient has read the information note and signed the informed consent form.
* The patient is covered by social security.

Exclusion Criteria:

* Patient age < 18 years
* Patients diagnosed with metastatic or bilateral breast cancer
* Patients with metastatic disease of any location
* Peripheral neuropathy grade ≥ 2 according to CTCAE version 5.0 of the upper or lower limbs
* Patients with asymmetric upper limb peripheral neuropathy grade > 1 according to CTCAE version 5.0 at inclusion.

  *In the case of asymmetry of the lower limbs of grade > 1 according to CTCAE version 5.0, the patient will not be considered a failure in selection but the corresponding secondary criteria will not be analysed.
* Patients with underlying medical conditions that could potentially cause peripheral neuropathy (diabetes mellitus, chronic alcoholism, unilateral lymphoedema or postherpetic neuralgia), or any other reason based on the investigator's judgement.
* Diagnosed Raynaud's syndrome
* Obstructive arterial disease of the lower limbs
* History of myocardial infarction
* Patients already using compression foot socks
* Vulnerable populations and participants defined in Articles 64 to 68 of Regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017:

  * Pregnant women
  * Incapacitated participants who have not given their free and informed consent or refused to do so before the onset of their incapacity, who do not fall under the provisions of Article 64 ;
  * Pregnant or breast-feeding women who are not covered by the provisions of article 66;
  * Persons of full age who are the subject of a legal protection measure or who are unable to express their consent.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy in preventing peripheral neuropathy as determined by medical staff between cryotherapy treatment alone and combined cryotherapy and compression treatment of the upper limbs in patients treated with paclitaxel. | 7 days after completion of C3D15 or C4D1 if applicable (each cycle is 21 days)
  The limb with the highest grade of neuropathy will be given a score of 1 and the limb with the lowest grade of neuropathy a score of 0. If no neuropathy is identified in either of the 2 limbs, a score of 0 will be given for each limb. Finally, if a neuropathy of the same grade is identified in each of the 2 limbs, a score of 1 will be assigned for both limbs.
  Success is defined as a differential of -1 in neuropathy score in favour of double prevention. This method will be applied to the primary and secondary endpoints.

SECONDARY OUTCOMES:
To compare the efficacy of cryotherapy alone and combined cryotherapy and compression treatment of the upper limbs in reducing the occurrence of peripheral neuropathy as determined by medical staff throughout the course of treatment. | At inclusion, just before each treatment cycle (C1D1, C2D1, C3D1) (each cycle is 21 days), at 1 month (±2 weeks) and at 4 months after the end of chemotherapy (±2 weeks)
  Differential between the two upper limbs
To compare the efficacy of cryotherapy alone and combined cryotherapy and compression treatment of the lower limbs in reducing the occurrence of peripheral neuropathy as determined by medical staff throughout the course of treatment. | At inclusion, just before each treatment cycle (C1D1, C2D1, C3D1 and 7 days after C3D15 or C4D1 if applicable), (each cycle is 21 days) at 1 month (±2 weeks) and at 4 months after the end of chemotherapy (±2 weeks)
  Differential between the two upper limbs
To compare the efficacy of cryotherapy alone and combined cryotherapy and compression treatment of the lower limbs in reducing the occurrence of peripheral neuropathy as determined by the patient throughout the course of treatment. | At inclusion, just before each treatment cycle (C1D1, C2D1, C3D1 and 7 days after C3D15 or C4D1 if applicable) (each cycle is 21 days), at 1 month (±2 weeks) and at 4 months after the end of chemotherapy (±2 weeks)
  Differential between the two lower limbs
Comparing cryotherapy tolerance rates with and without compression | During D1, D8 and D15 of all cycles ((each cycle is 21 days)
  Rate of discontinuation of cryotherapy during treatment
Evaluate the impact of compression on the temperature at the extremities | 15 minutes before and after removal of cryotherapy and compression devices at D1, D8 and D15 of each chemotherapy cycle (each cycle is 21 days)
  Comparison of the temperature measured between the upper and lower limbs (at extremity level) using an infrared thermometer
Study the percentage and characteristics of peripheral neuropathy according to the DN4 questionnaire during treatment | C1D1, C2D1, C3D1 and 7 days after C3D15), (each cycle is 21 days) at 1 month (±2 weeks) and 4 months after the end of chemotherapy (±2 weeks).
  Percentage of patients with peripheral neuropathy for any limb according to the results of the DN4 questionnaire just before each treatment cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No